CLINICAL TRIAL: NCT06430632
Title: Early Robotic Gait Training After Stroke
Acronym: ERA Stroke
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Baylor Research Institute (Other)
Collaborators: National Institute on Disability, Independent Living, and Rehabilitation Research (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 023-471; 90IFRE0074 (Other Grant/Funding Number: National Institute on Disability, Independent Living, and Rehabilitation Research)
Record Dates: First submitted 2024-05-09; First posted 2024-05-28 (Actual); Last update posted 2026-02-06 (Actual); Status verified 2026-02

CONDITIONS: Stroke
Keywords: Exoskeleton; Gait training; Inpatient rehabilitation; Physical therapy; Physical rehabilitation and medicine; Randomized controlled trial; Robotic gait training
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Intervention Model Description: Participants will be randomized to either the experimental group receiving robotic gait training or the control group receiving usual care gait training.
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Robotic Gait Training (Experimental): Participants will receive robotic gait training with a physical therapist for 90 minutes each week throughout the course of their inpatient rehabilitation stay.
  Interventions: Device: Robotic Gait Training
- Usual Care Gait Training (Active Comparator): Participants will receive usual care gait training with a physical therapist for 90 minutes each week throughout the course of their inpatient rehabilitation stay.
  Interventions: Other: Usual Care Gait Training

INTERVENTIONS:
Device: Robotic Gait Training — Participants will complete standing and walking activities while wearing a robotic exoskeleton. Participants will also be asked to complete questionnaires about their walking and function.
  Other Names: EksoNR Robotic Exoskeleton
  Arms: Robotic Gait Training
Other: Usual Care Gait Training — Participants will complete standing and walking activities such as body weight-supported treadmill training and conventional overground walking. Participants will also be asked to complete questionnaires about their walking and function.
  Other Names: Standard of Care Gait Training
  Arms: Usual Care Gait Training

SUMMARY:
The ERA Stroke project will compare the effects of robotic gait training (RGT) and usual care (UC) gait training in patients in the subacute phase of stroke recovery undergoing inpatient rehabilitation at the Baylor Scott & White Institute for Rehabilitation (BSWIR).

DETAILED DESCRIPTION:
Importance: Stroke is estimated to affect 6.6 million Americans, and around 795,000 new cases are reported each year. By 2030, annual stroke-related healthcare costs are expected to eclipse $240 billion, a staggering 445% increase from the current annual cost of $53.9 billion. Specialized stroke rehabilitation reduces long-term disability and stroke-related costs, making cost-efficient efforts to minimize functional deficits faced by people with stroke (e.g., gait impairment) a high priority. This project will provision preliminary evidence regarding the clinical use and efficacy of robotic gait training (RGT) during the subacute phase of stroke recovery as well as observational findings associated with the safety, tolerability, feasibility, and cost of delivering RGT during inpatient stroke rehabilitation. Its results will help with developing safe, tolerable, and cost-effective training protocols to improve walking function after stroke. Additionally, follow-up assessments after discharge will investigate any carryover effect of RGT, providing foundational data to evaluate the dose-response relationship for delivering RGT during inpatient rehabilitation after stroke. Altogether, this evidence will help stroke rehabilitation programs to assess their planning and budgeting needs prior to adopting RGT technology, improving outcomes and lowering lifetime care costs for patients with stroke.

Aims: (1) Evaluate the safety, tolerability, and feasibility of delivering an RGT intervention that meets the unique needs of people after stroke during inpatient rehabilitation informed by an Advisory Board comprised of stakeholders living with stroke. (2) Examine the efficacy of RGT compared to usual care (UC) gait training during inpatient rehabilitation for people with stroke. (3) Conduct a cost analysis of delivering RGT during inpatient rehabilitation compared to UC.

Methods: This randomized controlled trial will enroll 54 patients admitted to the Baylor Scott and White Institute for Rehabilitation following stroke. Participants will be randomized to either the experimental group receiving RGT or the control group receiving UC.

Addition to State-of-the-Art: Expected products include a manualized, stakeholder-informed RGT intervention and cost-analysis template that can be replicated across early rehabilitation settings nationally for people with stroke.

Sustained Approach: This project builds upon our earlier findings to achieve optimal walking recovery post-stroke during inpatient rehabilitation. The proposed work will generate preliminary efficacy, safety, tolerability, feasibility, and cost-analysis data concerning delivering an RGT intervention during the subacute phase for people with stroke.

ELIGIBILITY:
Inclusion Criteria:

* 18-85 years of age
* All types of stroke
* Acute/subacute phase of recovery
* Medically stable as deemed by a physician
* Undergoing medical care and rehabilitation at BSWIR
* All genders, races, and ethnicities
* Meets Ekso robotic exoskeleton frame limitations
* Continence or on a program for bladder and bowel management
* Capacity and goal for walking recovery

Exclusion Criteria:

* Concurrent neurological diagnoses (e.g., TBI, degenerative, CNS neoplasm)
* Profound cognitive impairment
* Pregnancy

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 54 (Estimated)
Dates: Start 2024-03-01 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Gait speed via 10-Meter Walk Test (10MWT) | within 7 days of admission to inpatient rehabilitation, within 7 days of discharge from inpatient rehabilitation, 1 month (±14 days) after discharge from inpatient rehabilitation, 3 months (±14 days) after discharge from inpatient rehabilitation
  The 10MWT assesses gait speed over a short duration. Gait speed (m/s) is correlated with ability to mobilize in the community, capacity to perform activities of daily living, and risk of falls, re-hospitalization, and cognitive decline. The 10MWT can be used to categorize individuals according to their ambulatory ability: household ambulators (<0.4 m/s), limited community ambulators (0.4 to 0.8 m/s), and community ambulators (>0.8 m/s). Score changes >0.16 m/s exceed the MCID. Normal gait speed for adults older than 50 years is >1.27 m/s.

SECONDARY OUTCOMES:
Functional Ambulation Category (FAC) | within 7 days of admission to inpatient rehabilitation, within 7 days of discharge from inpatient rehabilitation, 1 month (±14 days) after discharge from inpatient rehabilitation, 3 months (±14 days) after discharge from inpatient rehabilitation
  The FAC assesses functional ambulation in patients undergoing rehabilitation and has excellent reliability, good predictive validity, and good responsiveness in patients with stroke. Scores range from 0 (unable to walk) to 5 (independent walking anywhere). After 4 weeks of rehabilitation, FAC scores ≥4 predict community ambulation at 6 months with 100% sensitivity and 78% specificity.
Continuity Assessment Record and Evaluation (CARE) | within 7 days of admission to inpatient rehabilitation, within 7 days of discharge from inpatient rehabilitation, 1 month (±14 days) after discharge from inpatient rehabilitation, 3 months (±14 days) after discharge from inpatient rehabilitation
  The Section GG CARE is utilized in post-acute care settings for tracking progress across the continuum of care and is conducted at admission and discharge. The CARE addresses self-care (GG0130, 8 items) and functional mobility (GG0170, 17 items). Scores for each item range from 1 (dependent) to 6 (independent). Total scores for the CARE have strong positive correlations with total scores for the Functional Independence Measure.
6-Minute Walk Test (6MWT) | within 7 days of admission to inpatient rehabilitation, within 7 days of discharge from inpatient rehabilitation, 1 month (±14 days) after discharge from inpatient rehabilitation, 3 months (±14 days) after discharge from inpatient rehabilitation
  The 6MWT assesses distance walked over 6 minutes as a sub-maximal test of walking capacity. Endurance (captured as walking capacity) is essential to participate in community-based activities. With excellent test-retest reliability (ICC = 0.99) for people with stroke, the established MCID is 34.4 meters.
Modified Rankin Scale (mRS) | within 7 days of admission to inpatient rehabilitation, within 7 days of discharge from inpatient rehabilitation, 1 month (±14 days) after discharge from inpatient rehabilitation, 3 months (±14 days) after discharge from inpatient rehabilitation
  The mRS measures the degree of disability or dependence in the daily activities of people who have had a stroke. The mRS is an ordinal scale with 6 categories ranging from 0 (no symptoms) to 5 (complete physical dependence).
Stroke Rehabilitation Assessment of Movement (STREAM) | within 7 days of admission to inpatient rehabilitation, within 7 days of discharge from inpatient rehabilitation, 1 month (±14 days) after discharge from inpatient rehabilitation, 3 months (±14 days) after discharge from inpatient rehabilitation
  The STREAM assesses upper and lower limb motor function along with basic mobility in people with stroke and has a very high inter-rater reliability (ICC = 0.96). MCID values have been established for the upper extremity (2.2 points), lower extremity (1.9 points), and mobility (4.8 points) subscales.
5 Times Sit-to-Stand Test (5TSST) | within 7 days of admission to inpatient rehabilitation, within 7 days of discharge from inpatient rehabilitation, 1 month (±14 days) after discharge from inpatient rehabilitation, 3 months (±14 days) after discharge from inpatient rehabilitation
  The 5TSST assesses lower extremity strength and is an indicator of postural control. People with stroke who score >15 seconds are considered at risk for falls. Normal scores for individuals aged 60-80 years range from 11.4 to 12.7 seconds. The 5TSST has demonstrated excellent test-retest reliability (ICC = 0.95) with an established MDC95 of 2.3 seconds.
Berg Balance Scale (BBS) | within 7 days of admission to inpatient rehabilitation, within 7 days of discharge from inpatient rehabilitation, 1 month (±14 days) after discharge from inpatient rehabilitation, 3 months (±14 days) after discharge from inpatient rehabilitation
  The BBS is a 14-item objective measure that assesses static balance and fall risk in adults. With excellent reliability (ICC = 0.95), the BBS has a large responsiveness for acute stroke (effect size = 0.85) and a minimal detectable change of 6.9 points. Scores <45/56 indicate a risk of falling.
Stroke Impact Scale - 16 (SIS-16) | within 7 days of admission to inpatient rehabilitation, within 7 days of discharge from inpatient rehabilitation, 1 month (±14 days) after discharge from inpatient rehabilitation, 3 months (±14 days) after discharge from inpatient rehabilitation
  The SIS-16 assesses 4 dimensions of health-related QOLs specific to people who have had a stroke. It includes subscales that assess strength, hand function, mobility, and activities of daily living via 5-point Likert scales.
Rating of Perceived Exertion (RPE) | immediately following every treatment session until discharge from inpatient rehabilitation (an average of 2 weeks)
  The Borg RPE is a 15-point scale with verbal descriptors to standardize perceived exertion across tasks and individuals. Participants will be asked to provide a self-reported intensity level on the Borg Rating of Perceived Exertion Scale during RGT and UC gait training sessions. A self-report of 12 to 14 on the RPE indicates moderate intensity.
Number of steps (RGT only) | immediately following every treatment session until discharge from inpatient rehabilitation (an average of 2 weeks)
  The Ekso device records several data points for each session including number of steps, "Up" time (the amount of time spent standing in the device), "Walk" time (the amount of time spent walking in the device), and device assistance scores. While all of these data values will be recorded to describe each RGT session and tracked to monitor progression of the RGT intervention, the number of steps per session will be utilized as an indicator of RGT session intensity.
Distance walked (UC only) | immediately following every treatment session until discharge from inpatient rehabilitation (an average of 2 weeks)
  Distance walked will be recorded to describe each UC session, tracked to monitor progression of the UC intervention, and utilized as an indicator of UC session intensity.

OTHER OUTCOMES:
Gait quality | weekly until discharge from inpatient rehabilitation (an average of 2 weeks)
  To supplement the study's measurements of RGT efficacy (10-meter walk test [gait speed], 6-minute walk test [gait endurance], and Functional Ambulation Category [gait independence]), the investigators will additionally measure gait quality. Improvements in quality of gait after a stroke are associated with gains in balance and functional mobility. Further, return to participation in life roles is largely associated with a patients' perspective on their recovery. Therefore, the most impactful way to capture gait quality for each participant will be to use a measure of self-report. Specifically, gait quality will be measured weekly on a visual analog scale from 1 ("my walking is the worst it has ever been") to 10 ("my walking is just like before my stroke").
Pain following each gait training session | weekly until discharge from inpatient rehabilitation (an average of 2 weeks)
  Pain after stroke is common and can result in reduced participation in activity. This change will allow the investigators to monitor the impact of pain on gait outcomes. Pain will be assessed following each RGT and UC session using a pain visual analog scale, as per standard of care in the investigators' inpatient rehabilitation hospital.
Adverse event rate | through study completion (up to 3.5 months)
  Number of adverse events occurring at baseline through study completion.
Treatment tolerability (RGT only) | weekly until discharge from inpatient rehabilitation (an average of 2 weeks)
  Subjects will provide feedback on their tolerance of treatment sessions via a questionnaire that measures tolerability on a scale 0 (not tolerable at all) to 10 (maximally tolerable). A higher score means greater tolerability in robotic gait training.
Treatment completion rate | through study completion (up to 3.5 months)
  The number of sessions attended divided by the number of scheduled sessions.

CONTACTS AND LOCATIONS:
Locations (1):
- Baylor Scott & White Institute for Rehabilitation, Dallas, Texas, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] da Silva Areas FZ, Baltz S, Gillespie J, Ochoa C, Gilliland T, Dubiel R, Bennett M, Driver S, Swank C. Early robotic gait training after stroke (ERA Stroke): study protocol for a randomized clinical trial. BMC Neurol. 2024 Oct 18;24(1):401. doi: 10.1186/s12883-024-03858-y. PMID 39425088